CLINICAL TRIAL: NCT01241448
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2b Study of LY2409021 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY2409021 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13031; I1R-MC-GLBG (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — adomeglivant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Taken orally once daily for 24 weeks. Participants who entered the study on stable metformin therapy were to continue at the dose prescribed by their physician.
  Interventions: Drug: Placebo
- 2.5 mg LY2409021 (Experimental): Taken orally once daily for 24 weeks. Participants who entered the study on stable metformin therapy were to continue at the dose prescribed by their physician.
  Interventions: Drug: LY2409021
- 10 mg LY2409021 (Experimental): Taken orally once daily for 24 weeks. Participants who entered the study on stable metformin therapy were to continue at the dose prescribed by their physician.
  Interventions: Drug: LY2409021
- 20 mg LY2409021 (Experimental): Taken orally once daily for 24 weeks. Participants who entered the study on stable metformin therapy were to continue at the dose prescribed by their physician.
  Interventions: Drug: LY2409021

INTERVENTIONS:
Drug: LY2409021 — Administered Orally
  Arms: 10 mg LY2409021; 2.5 mg LY2409021; 20 mg LY2409021
Drug: Placebo — Administered Orally
  Arms: Placebo

SUMMARY:
LY2409021 is being evaluated for possible treatment in type 2 diabetes. This study is designed to compare LY2409021 given alone or given in combination with metformin against placebo the change in hemoglobin A1c after a 24-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Type 2 diabetes mellitus according to the World Health Organization (WHO) diagnostic criteria
* Are women not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause.
* Are male patients using a reliable method of birth control during the study and until 3 months after the last dose of study medication.
* Are being treated with either diet and exercise alone, or with diet and exercise in combination with metformin. Metformin therapy must have been stable and unchanged for at least 3 months prior to screening and at a dose of at least 1000 milligram per day (mg/day).
* Have a hemoglobin A1c (HbA1c) value of 7.0% to 10.5%, inclusive.
* Have a body mass index (BMI) between 25 to 45 kilogram per meter squared (kg/m^2), inclusive.

In the opinion of the investigator, are capable and willing to:

* Perform self-monitoring of blood glucose
* Complete a study diary as required for this protocol
* Maintain consistent dietary, physical activity, and sleeping patterns throughout the duration of the study
* Comply with treatment regimens
* Have given written informed consent to participate in this study in accordance with local regulations and the Ethical Review Board (ERB) governing the study site.

Exclusion Criteria:

* Have more than 1 episode of severe hypoglycemia (defined as an event during which the patient requires the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions) within 6 months prior to screening, or have a current diagnosis of hypoglycemia unawareness.
* Have had two or more emergency room visits or hospitalizations due to poor glucose control in the 6 months prior to screening.
* Have gastrointestinal disease that may significantly impact gastric emptying or motility or have undergone gastric bypass or gastric banding surgery.
* Have had a previous diagnosis of pancreatitis.
* Have New York Heart Association (NYHA) class II, III, or IV symptoms of heart failure
* Have a history of myocardial infarction, unstable angina, or a coronary revascularization procedure within 6 months of screening.
* Have a history of supraventricular tachycardia, ventricular tachycardia, or other cardiac arrhythmia.
* Have a history of transient ischemic attack (TIA) or stroke within 6 months of screening.
* Have poorly controlled hypertension (systolic blood pressure greater than or equal to 150 mm Hg or diastolic blood pressure greater than or equal to 90 mm Hg) as determined by the mean of three separate measurements.
* Show evidence of labile blood pressure, including symptomatic postural hypotension.
* Have any abnormality of the ECG that would impact patient safety or data interpretation.
* Show clinical signs or symptoms of liver disease, or liver function tests (LFTs; aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) greater than 2.5 times upper limit of normal (ULN) as determined by the central laboratory at screening.
* Have a current or previous diagnosis of Gilbert's disease.
* Have previous or current diagnosis of Hepatitis B or C
* Have a serum creatinine >2 milligrams per deciliter (mg/dL) or, in patients being treated with metformin, a serum creatinine above (or creatinine clearance below) what is approved in the metformin product labeling in the respective country.
* Show evidence of uncorrected hypothyroidism or hyperthyroidism based on clinical evaluation and/or an abnormal thyroid stimulating hormone result as determined by the central laboratory at screening; patients receiving dose-stable thyroid replacement therapy for at least 3 months prior to screening will be allowed to participate in the study.
* Have any other abnormal laboratory value that, in the opinion of the investigator, precludes the patient from participation in the study. Laboratory abnormalities consistent with type 2 diabetes mellitus and all other eligibility criteria are acceptable: for example, abnormalities of blood glucose, hemoglobin A1c (HbA1c), urinary glucose, and urinary protein (with a range of trace to 1+ on dipstick).
* Have a currently suspected or treated malignancy, or are in remission from a clinically significant malignancy (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years.
* Have a personal or family history of pancreatic neoplasia.
* Have non-fasting triglycerides >600 mg/dL.
* Use or have used insulin or GLP-1 agonists (for more than 1 week within the 3-month period prior to screening), or any oral antihyperglycemic medication (OAM) other than metformin within the 3-month period prior to screening.
* Currently use or intend to use prescription or over-the-counter medications, including herbal supplements, to promote weight loss or to regulate blood glucose.
* Have current chronic (>2 weeks) systemic glucocorticoid therapy (excluding ocular topical, other topical, inhaled preparations) or have received such therapy within 8 weeks prior to screening.
* Currently use hyperglycemia-causing agents, hypoglycemia-causing agents (other than metformin), class II and III antiarrythmic agents, agents that reduce gastrointestinal motility, central nervous system stimulants (with the exception of caffeinated beverages), fibrates, and niacin greater than or equal to 1 grams per day (gm/day).
* Have an average weekly alcohol intake that exceeds 2 units per day for males and 1 unit per day for females (1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 milliliters (mL) of wine; 1.5 oz or 45 milliliter (mL) of distilled spirits).
* Currently use drugs with a narrow therapeutic index (for example, digoxin, lithium, phenytoin, theophylline, and warfarin).
* Currently use drugs that are known to prolong the QT interval.
* Currently use or intend to use potent inhibitors of CYP3A, which include but are not limited to atazanavir, indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone, saquinavir, and telithromycin.
* Have previously completed or withdrawn from this study or any other study investigating LY2409021.
* Have known allergies to LY2409021 or related compounds.
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or unapproved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have any other condition such as alcohol abuse, drug abuse, or psychiatric disorder that may affect the ability to participate in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-4559) or 1-317-615-4559 Mon - Fri 9 Am - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (40):
- United States (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burbank, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mission Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Springs, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roseville, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Luis Obispo, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meridian, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Henderson, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilmington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Damme
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elsterwerda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., HohenmÃ¶lsen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., LÃ¼neburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ludwigshafen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chieti Scalo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hato Rey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Romania (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- Slovakia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Košice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Malacky
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville

REFERENCES:
- [Derived] Kazda CM, Ding Y, Kelly RP, Garhyan P, Shi C, Lim CN, Fu H, Watson DE, Lewin AJ, Landschulz WH, Deeg MA, Moller DE, Hardy TA. Evaluation of Efficacy and Safety of the Glucagon Receptor Antagonist LY2409021 in Patients With Type 2 Diabetes: 12- and 24-Week Phase 2 Studies. Diabetes Care. 2016 Jul;39(7):1241-9. doi: 10.2337/dc15-1643. Epub 2015 Dec 17. PMID 26681715

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo orally once daily for 24 weeks. Participants who entered the study on stable metformin therapy were to continue at the dose prescribed by their physician.
- 2.5 mg LY2409021: 2.5 mg LY2409021 orally once daily for 24 weeks. Participants who entered the study on stable metformin therapy were to continue at the dose prescribed by their physician.
- 10 mg LY2409021: 10 mg LY2409021 orally once daily for 24 weeks. Participants who entered the study on stable metformin therapy were to continue at the dose prescribed by their physician.
- 20 mg LY2409021: 20 mg LY2409021 orally once daily for 24 weeks. Participants who entered the study on stable metformin therapy were to continue at the dose prescribed by their physician.
Period: Overall Study
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Started | 66 | 65 | 66 | 66
Intent-to-Treat Population (ITT) | 63 | 63 | 64 | 64
ITT With ≥1 Post-Baseline Measure | 61 | 61 | 64 | 62
Completed | 29 | 36 | 43 | 43
Not Completed | 37 | 29 | 23 | 23
Not completed — Adverse Event | 1 | 0 | 2 | 2
Not completed — Lost to Follow-up | 2 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 10 | 5 | 3 | 6
Not completed — Sponsor Decision | 17 | 14 | 12 | 6
Not completed — Withdrawal by Subject | 4 | 5 | 3 | 6
Not completed — Excluded due to data integrity issues | 3 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline data is provided for all randomized participants excluding the 9 participants from a single site where data integrity issues were identified (Intent-to-treat population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021 | Total
Number analyzed (Participants) | 63 | 63 | 64 | 64 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (8.79) | 57.3 (8.23) | 54.6 (8.05) | 55.9 (8.82) | 55.7 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 17 | 19 | 83
  Male | 40 | 39 | 47 | 45 | 171
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 25 | 26 | 28 | 108
  Slovakia | 7 | 7 | 6 | 6 | 26
  Puerto Rico | 3 | 4 | 3 | 5 | 15
  Spain | 6 | 7 | 7 | 7 | 27
  Romania | 10 | 12 | 12 | 10 | 44
  Germany | 7 | 7 | 9 | 6 | 29
  Italy | 1 | 1 | 1 | 2 | 5
Race [Count of Participants; unit: Participants]
  Asian | 1 | 3 | 1 | 0 | 5
  Black or African American | 4 | 6 | 2 | 6 | 18
  White | 58 | 54 | 61 | 58 | 231
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 14 | 13 | 13 | 56
  Not Hispanic or Latino | 36 | 31 | 35 | 37 | 139
  Not Reported | 11 | 18 | 16 | 14 | 59
Diabetes Duration [Mean (Standard Deviation); unit: years] | 5.8 (5.29) | 6.9 (7.23) | 5.5 (4.21) | 5.8 (6.13) | 6.0 (5.81)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m^2)] | 32.1 (4.63) | 31.9 (4.86) | 32.3 (4.91) | 32.6 (5.27) | 32.2 (4.90)
Waist Circumference [Mean (Standard Deviation); unit: centimeters (cm)] | 106.7 (12.41) | 107.5 (11.16) | 107.2 (12.24) | 106.8 (12.28) | 107.1 (11.97)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of Hemoglobin A1c (HbA1c)] | 8.1 (1.00) | 8.1 (0.93) | 8.1 (0.87) | 8.0 (0.92) | 8.0 (0.92)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 24 Week Endpoint in Hemoglobin A1c (HbA1c)
Description: Least squares means of the change from baseline is from a mixed-model repeated measures analysis (MMRM). The model included terms for treatment group, baseline HbA1c, metformin use, visit, and visit-by-treatment interaction.
Time Frame: Baseline, 24 weeks
Population: All participants randomly assigned to treatment with at least 1 post-baseline HbA1c measurement (excluding participant data from the excluded site); analyzed according to the treatment to which the participants were randomly assigned.
Measure: Least Squares Mean (90% Confidence Interval); unit: percentage of Hemoglobin A1c (HbA1c)
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 61 | 61 | 63 | 60
percentage of Hemoglobin A1c (HbA1c) | -0.15 [-0.37 to 0.06] | -0.45 [-0.65 to -0.25] | -0.78 [-0.97 to -0.58] | -0.92 [-1.12 to -0.73]
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg LY2409021; Sixty-five randomized patients (45 completers) per arm were expected to provide at least 90% power to detect 0.8% HbA1c difference with placebo assuming a SD for change in HbA1c of 1.2% (0.05 1-sided type I error); Test type: Superiority or Other; p = 0.094, Mixed Models Analysis — No multiplicity adjustments were used to calculate the p-value; Least Squares Mean Difference = -0.29, 90% CI 2-sided [-0.58 to -0.01]
Statistical Analysis 2: Comparison: Placebo vs 10 mg LY2409021; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — No multiplicity adjustments were used to calculate the p-value; Least Squares Mean Difference = -0.62, 90% CI 2-sided [-0.90 to -0.34]
Statistical Analysis 3: Comparison: Placebo vs 20 mg LY2409021; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis — No multiplicity adjustments were used to calculate the p-value; Least Squares Mean Difference = -0.77, 90% CI 2-sided [-1.05 to -0.48]

2. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Fasting Blood Glucose (FBG)
Description: Least squares means of the change from baseline is from a mixed-model repeated measures analysis (MMRM). The model included terms for treatment group, baseline value, metformin use, visit, and visit-by-treatment interaction.
Time Frame: Baseline, 24 weeks
Population: All participants randomly assigned to treatment with at least 1 post-baseline laboratory FBG measurement (excluding participant data from the excluded site); analyzed according to the treatment to which the patients were randomly assigned.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 60 | 59 | 62 | 60
millimoles per liter (mmol/L) | -0.36 [-0.92 to 0.21] | -0.46 [-0.99 to 0.07] | -1.07 [-1.57 to -0.56] | -1.14 [-1.66 to -0.62]

3. Secondary Outcome: Change From Baseline to 24 Week Endpoint in 7-point Self Monitored Glucose (SMBG) Profile
Description: SMBG profiles consisted of blood glucose values collected before and 2 hours after the 3 main meals and at 0300 hours (3:00 AM). Values represent mean of values collected same time on 3 separate days within a week prior to visit. Least squares (LS) mean of the change from baseline is from a mixed-model repeated measures analysis (MMRM). The model included terms for treatment group, baseline value, metformin use, visit, and visit-by-treatment interaction.
Time Frame: Baseline, 24 weeks
Population: All randomized patients with at least 1 post-baseline self-monitored glucose measurement (excluding participant data from the excluded site); analyzed according to the treatment to which the patients were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 54 | 56 | 59 | 59
milligrams per deciliter (mg/dL)
  Pre-morning meal (fasting): number analyzed (Participants) | 54 | 55 | 58 | 59
  Pre-morning meal (fasting) | -14.45 [-22.26 to -6.63] | -15.76 [-22.78 to -8.74] | -29.65 [-36.56 to -22.73] | -32.55 [-39.46 to -25.64]
  2 hours after morning meal: number analyzed (Participants) | 54 | 55 | 58 | 59
  2 hours after morning meal | -28.75 [-39.55 to -17.95] | -23.01 [-32.66 to -13.35] | -48.12 [-57.42 to -38.83] | -45.76 [-55.05 to -36.47]
  Pre-mid-day meal: number analyzed (Participants) | 54 | 54 | 58 | 59
  Pre-mid-day meal | -17.83 [-27.33 to -8.33] | -16.13 [-24.66 to -7.61] | -27.35 [-35.49 to -19.20] | -25.45 [-33.66 to -17.24]
  2 hours after mid-day meal: number analyzed (Participants) | 53 | 54 | 58 | 58
  2 hours after mid-day meal | -23.75 [-34.61 to -12.89] | -21.17 [-30.75 to -11.58] | -31.42 [-40.70 to -22.14] | -39.60 [-49.01 to -30.19]
  Pre-evening meal: number analyzed (Participants) | 53 | 55 | 58 | 59
  Pre-evening meal | -7.45 [-18.88 to 3.98] | -11.77 [-21.87 to -1.66] | -14.15 [-23.95 to -4.36] | -25.02 [-34.82 to -15.22]
  2 hours after evening meal: number analyzed (Participants) | 54 | 54 | 58 | 59
  2 hours after evening meal | -19.48 [-30.67 to -8.30] | -21.74 [-31.67 to -11.81] | -33.93 [-43.42 to -24.45] | -32.01 [-41.53 to -22.49]
  0300 hours (3:00 AM): number analyzed (Participants) | 54 | 47 | 55 | 54
  0300 hours (3:00 AM) | -5.13 [-14.77 to 4.50] | -9.52 [-18.59 to -0.45] | -23.33 [-31.74 to -14.91] | -25.67 [-34.44 to -16.89]

4. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Plasma Glucose
Description: as for outcome 2
Time Frame: Baseline, 24 weeks
Population: All randomized patients with at least 1 post-baseline plasma glucose measurement (excluding participant data from the excluded site); analyzed according to the treatment to which the patients were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 60 | 59 | 62 | 60
millimoles per liter (mmol/L) | -0.36 [-0.92 to 0.21] | -0.46 [-0.99 to 0.07] | -1.07 [-1.57 to -0.56] | -1.14 [-1.66 to -0.62]

5. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Fasting Insulin
Description: Least squares (LS) mean of the change from baseline is from a mixed-model repeated measures analysis (MMRM). The model included terms for treatment group, baseline value, metformin use, visit, and visit-by-treatment interaction.
Time Frame: Baseline, 24 weeks
Population: All randomized patients with at least 1 post-baseline fasting insulin measurement (excluding participant data from the excluded site); analyzed according to the treatment to which the patients were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: picomoles per liter (pmol/L)
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 55 | 58 | 60 | 59
picomoles per liter (pmol/L) | 10.62 [-3.87 to 25.11] | 2.61 [-9.77 to 14.98] | 14.95 [3.54 to 26.36] | 9.65 [-2.56 to 21.87]

6. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Fasting Glucagon-like Peptide 1 (GLP-1) Active and Total
Description: GLP-1 is cleaved from proglucagon to form the active peptide GLP-1. The active form promotes suppression of glucagon secretion. Total GLP-1 is the active GLP-1 and the Dipeptidyl Peptidase IV cleaved GLP-1 form. Least squares (LS) mean of the change from baseline is from a mixed-model repeated measures analysis (MMRM). The model included terms for treatment group, baseline value, metformin use, visit, and visit-by-treatment interaction.
Time Frame: Baseline, 24 weeks
Population: All randomized patients with at least 1 post-baseline GLP-1 active and total measurements (excluding participant data from the excluded site); analyzed according to the treatment to which the patients were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: picomoles per liter (pmol/L)
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 56 | 58 | 62 | 59
picomoles per liter (pmol/L)
  Active GLP-1 | -0.30 [-0.88 to 0.28] | 0.13 [-0.40 to 0.66] | 0.38 [-0.11 to 0.87] | 0.31 [-0.20 to 0.82]
  Total GLP-1: number analyzed (Participants) | 55 | 58 | 62 | 59
  Total GLP-1 | -0.12 [-1.50 to 1.27] | 1.84 [0.60 to 3.08] | 4.63 [3.48 to 5.79] | 8.23 [7.04 to 9.42]

7. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Fasting Lipid Profile
Description: Fasting Lipid Profile included: Triglycerides, Low Density Lipoprotein Cholesterol (LDL-C), High Density Lipoprotein Cholesterol (HDL-C) and Total Cholesterol. Least squares (LS) mean of the change from baseline is from a mixed-model repeated measures analysis (MMRM). The model included terms for treatment group, baseline value, visit, and visit-by-treatment interaction.
Time Frame: Baseline, 24 weeks
Population: All randomized patients with at least 1 post-baseline fasting lipid measurement (excluding participant data from the excluded site); analyzed according to the treatment to which the patients were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 56 | 59 | 62 | 59
millimoles per liter (mmol/L)
  Triglycerides: number analyzed (Participants) | 50 | 53 | 58 | 55
  Triglycerides | -0.11 [-0.37 to 0.16] | 0.07 [-0.18 to 0.31] | 0.06 [-0.16 to 0.29] | 0.08 [-0.14 to 0.31]
  LDL-C: number analyzed (Participants) | 49 | 52 | 58 | 55
  LDL-C | 0.20 [-0.01 to 0.41] | 0.05 [-0.15 to 0.24] | 0.02 [-0.16 to 0.20] | 0.10 [-0.08 to 0.28]
  HDL-C: number analyzed (Participants) | 50 | 53 | 58 | 55
  HDL-C | 0.03 [-0.03 to 0.08] | 0.02 [-0.04 to 0.07] | 0.05 [0.00 to 0.10] | 0.04 [-0.01 to 0.09]
  Total Cholesterol: number analyzed (Participants) | 50 | 53 | 58 | 55
  Total Cholesterol | 0.15 [-0.08 to 0.39] | 0.10 [-0.11 to 0.31] | 0.10 [-0.10 to 0.30] | 0.19 [-0.01 to 0.39]

8. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Lipoprotein Subfractions-Particles (Total)
Description: Subfraction included: Very Low Density Lipoprotein (VLDL) Total. Least squares mean use an analysis of covariance model. The model included baseline lipoprotein subfractions, metformin use and treatment.
Time Frame: Baseline, 24 weeks
Population: All randomized patients with at least 1 post-baseline lipoprotein subfractions measurement (excluding participant data from the excluded site); analyzed according to the treatment to which the patients were randomized, last observation carried forward (LOCF) principle was applied.
Measure: Least Squares Mean (Standard Error); unit: nanomoles per liter (nmol/L)
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 52 | 59 | 61 | 55
nanomoles per liter (nmol/L) | 1.90 (4.296) | 6.48 (4.048) | 0.07 (4.099) | 2.04 (4.328)

9. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Free Fatty Acids
Description: Least squares mean use an analysis of covariance model. The model included baseline free fatty acid, metformin use and treatment.
Time Frame: Baseline, 24 weeks
Population: All randomized patients with at least 1 post-baseline free fatty acid measurement (excluding participant data from the excluded site); analyzed according to the treatment to which the patients were randomized.
Measure: Least Squares Mean (Standard Error); unit: picomoles per liter (pmol/L)
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 51 | 56 | 60 | 56
picomoles per liter (pmol/L) | -0.04 (0.043) | -0.02 (0.040) | -0.15 (0.037) | -0.07 (0.040)

10. Secondary Outcome: Change From Baseline to 24 Week Endpoint Indices in Insulin Sensitivity Using Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: HOMA-IR is a computer model (based on HOMA2) which uses fasting plasma insulin and glucose concentrations to estimate insulin resistance (HOMA-IR) as a proportion reference population (normal young adults). The normal reference population with normal function was indexed to 1.0. Higher values indicate increased insulin resistance. Least squares means of the change from baseline is from a mixed-model repeated measures analysis (MMRM). The model included terms for treatment group, baseline value, metformin use, visit, and visit-by-treatment interaction.
Time Frame: Baseline, 24 weeks
Population: All randomized patients with at least 1 post-baseline HOMA-IR measurement (excluding participant data from the excluded site); analyzed according to the treatment to which the patients were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: proportion of normal reference populatio
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 52 | 57 | 54 | 55
proportion of normal reference populatio | 0.19 [-0.10 to 0.49] | 0.02 [-0.24 to 0.27] | 0.26 [0.02 to 0.50] | 0.19 [-0.07 to 0.44]

11. Secondary Outcome: Change From Baseline to 24 Week Endpoint Indices in Beta-cell Function Using HOMA-B
Description: HOMA-B is a computer model (based on HOMA-2) that uses fasting plasma insulin and glucose concentrations to estimate steady state pancreatic beta cell function (%B) as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100%. Higher values indicate greater beta cell function. Least squares (LS) mean of the change from baseline is from a mixed-model repeated measures analysis (MMRM). The model included terms for treatment group, baseline value, metformin use, visit, and visit-by-treatment interaction.
Time Frame: Baseline, 24 week
Population: All randomized patients with at least 1 post-baseline HOMA-B measurement (excluding participant data from the excluded site); analyzed according to the treatment to which the patients were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent of normal reference population
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 52 | 57 | 54 | 55
percent of normal reference population | 4.88 [-3.27 to 13.03] | 7.90 [0.71 to 15.09] | 17.69 [10.94 to 24.43] | 16.39 [9.19 to 23.59]

12. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Weight
Description: Least squares means were adjusted for baseline weight, metformin use, visit, treatment and visit by treatment interaction.
Time Frame: Baseline, 24 weeks
Population: All randomized patients with at least 1 post-baseline weight measurement (excluding participant data from the excluded site); analyzed according to the treatment to which the patients were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms (kg)
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 61 | 61 | 64 | 61
kilograms (kg) | -1.07 [-2.20 to 0.05] | -0.33 [-1.39 to 0.73] | 0.55 [-0.46 to 1.55] | 0.07 [-0.95 to 1.10]

13. Secondary Outcome: Population Pharmacokinetics: Apparent Clearance (CL/F) of LY2409021
Description: Population pharmacokinetic parameter apparent clearance (CL/F) is the apparent volume of the body fluid cleared of the drug per unit of time and was estimated by modeling of LY2409021 plasma concentration data from all LY2409021 groups.
Time Frame: Baseline up to 26 weeks
Population: All randomized patients who received at least 1 one dose of study drug (excluding participant data from the excluded site); analyzed according to the treatment to which the patients were randomized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/hr)
Groups:
- LY2409021: 2.5 mg, 10 mg or 20 mg LY2409021 taken orally once daily for 24 weeks
Arm/Group | LY2409021
Number analyzed (Participants) | 191
liters per hour (L/hr) | 0.486 (31.0)

14. Secondary Outcome: Population Pharmacokinetics: Apparent Volume of Distribution of LY2409021
Description: Population pharmacokinetic parameter, apparent volume of distribution (V/F) is a theoretical volume that a drug would have to occupy (if it were uniformly distributed), to provide the same concentration as it currently is in blood plasma. Apparent volume of distribution (V/F) was estimated by modeling of LY2409021 plasma concentration data from all LY2409021 groups.
Time Frame: Baseline up to 26 weeks
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)
Arm/Group | LY2409021
Number analyzed (Participants) | 191
liters (L) | 33.4 (23.9)

15. Secondary Outcome: The Percentage of Participants Experiencing a Hypoglycemic Episode
Description: A hypoglycemic episode is any event during which typical symptoms of hypoglycemia are observed or when the measured plasma glucose concentration is less than or equal to 70 milligrams per deciliter (mg/dL) [3.9 millimoles per liter (mmol/L)].
Time Frame: Baseline through 24 weeks
Population: All randomized participants who received at least 1 dose of study drug (excluding participant data from the excluded site).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 63 | 63 | 64 | 64
percentage of participants | 3.2 | 6.3 | 9.4 | 7.8

16. Secondary Outcome: The 30-Day Adjusted Rate of Hypoglycemic Episodes
Description: A hypoglycemic episode is any event during which typical symptoms of hypoglycemia are observed or when the measured plasma glucose concentration is less than or equal to 70 milligrams per deciliter (mg/dL) [3.9 millimoles per liter (mmol/L)]. 30-day adjusted rate=(total number of episodes between 2 time intervals/number of days between intervals) X 30 days. Outcome measure was not analyzed due to the limited number of hypoglycemic events observed.
Time Frame: Baseline through 24 weeks
Population: Outcome measure was not analyzed due to the limited number of hypoglycemic events observed; therefore zero participants were analyzed.
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | 2.5 mg LY2409021 | 10 mg LY2409021 | 20 mg LY2409021
Serious Adverse Events (participants affected / at risk) | 3/66 | 0/65 | 2/66 | 2/66
Other Adverse Events (participants affected / at risk) | 23/66 | 31/65 | 34/66 | 29/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=66) | 2.5 mg LY2409021 (N=65) | 10 mg LY2409021 (N=66) | 20 mg LY2409021 (N=66)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=66) | 2.5 mg LY2409021 (N=65) | 10 mg LY2409021 (N=66) | 20 mg LY2409021 (N=66)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Type ii hyperlipidaemia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Type v hyperlipidaemia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (5) | 0 (0) | 2 (6)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (2) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 4 (4) | 3 (3)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (4) | 7 (11) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 7 (9) | 2 (2)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Colonoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Free fatty acids increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 3 (6) | 3 (3)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intermediate density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Abnormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 2 (2) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (3) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cluster headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (4) | 4 (4) | 4 (5)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (4) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental implantation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plastic surgery to the face (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous insufficiency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days